CLINICAL TRIAL: NCT01006746
Title: Evaluation and Description of Mutual Influences Between Patient Training, Perception and Adoption of Home-Monitoring Technology
Brief Title: Observational Study of Patient Comprehension, Perception, Fears and Appreciation Following Home-Monitoring Implementation
Acronym: Educ@t
Status: Completed | Type: Observational
Sponsor: Biotronik France (Industry)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: HS050
Record Dates: First submitted 2009-11-01; First posted 2009-11-03 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Defibrillators; Tachycardia
Keywords: Remote monitoring; Defibrillators; Survey; Indication for ICD (primary and secondary prevention)
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICD patient and Home Monitoring: Patients primo implanted with ICD
  Interventions: Other: Remote monitoring by Home Monitoring system

INTERVENTIONS:
Other: Remote monitoring by Home Monitoring system — Standard of care completed with remote monitoring for ICD patients follow-up
  Other Names: ICD: Lumax family (single-chamber, dual-chamber and CRT ICDs); Transmitter: cardioMessenger II or CardioMessenger IIs

SUMMARY:
Describe the mutual influences between trainings realized in implantation centers, medico-technical knowledges, technical implementation, perception, fears and appreciation felt by the patients during Home Monitoring implementation.

DETAILED DESCRIPTION:
500 patients with an indication for ICD (primary and secondary prevention) will be included in the registry during a period of 12 months. For the survey, patients must answer two questionnaires.

The first one will assess the knowledges regarding Home-Monitoring which certainly depend on the time devoted to patient information during the implantation. This period of training is important and has a direct impact on the CardioMessenger use by the patient. Although the study is multicenter, the aim is not to evaluate or compare practices of each center for the information provided to patients. The objective is to find ways to improve this phase.

A second questionnaire was designed to observe the perception of Home-monitoring by the patient and thus to understand how this new technology is apprehended. This part is important because we must take in consideration patient point of view and expectations to improve care and offer new products or services.

A focus on patients' perception and appreciation may give a support to the elaboration of training and prevention strategies, the anticipation of the needs, and the improvement of the technology. All these improvements may eventually take part in the success of ICD treatment.

ELIGIBILITY:
Inclusion Criteria:

* Primo ICD implantation with Home-Monitoring system

Exclusion Criteria:

* NYHA Class IV
* Pregnant women or women who plan to become pregnant during the trial
* Patient whose medical situation is not stable
* Presence of psychiatric illness, depression, anxiety disorders
* Presence of any disease, other than patient's cardiac disease, associated with reduced likelihood of survival for the duration of the trial, e.g. cancer, uraemia (urea > 70mg/dl or creatinine >3mg/dl, liver failure, etc.
* Age < 18 years
* Patient unable to handle the CardioMessenger correctly
* The patient is not willing and able to comply with the protocol (i.e. unable to answer to the questionnaires)
* Change of residence expected during the study
* Participation in another clinical study
* Patient unwilling to sign patient informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in 46 french investigational sites (hospitals and private clinics)
Sampling Method: Non-Probability Sample
Enrollment: 571 (Actual)
Dates: Start 2009-02; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
At 1 month: evaluation of centers training, knowledges and constraints of Home Monitoring implementation. At 6 months follow-up: observe and describe the behavior, the perception, the fears and the appreciation degree linked to this new technology | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Laurent, Dr, Principal Investigator — CHU Dijon
Locations (1):
- CHU Le Bocage, Dijon, Dijon, France